CLINICAL TRIAL: NCT06993610
Title: A Phase 2, Multi-Center Study Consisting of a Randomized, Placebo-Controlled Period, Followed by an Open-Label Extension Period to Assess the Efficacy, Safety, and Tolerability of Tibulizumab in Adults With Hidradenitis Suppurativa
Brief Title: Tibulizumab Skin Healing and Inflammation Evaluation for Lasting Defense
Acronym: TibuSHIELD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zura Bio Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZB-106-HS-202; 2024-519736-17-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-19; First posted 2025-05-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: Hidradenitis Suppurativa; HS; Tibulizumab; Hidradenitis Suppurativa clinical response; HiSCR; Skin Diseases; Inflammatory Skin Disease; Chronic Skin Condition; Sweat Gland Disease; Skin Diseases Bacterial; Suppurative Hidradenitis; Hidradenitis; Acne; Acne inversa; Inversa
MeSH Terms: conditions — Hidradenitis Suppurativa; Skin Diseases; Dermatitis; Sweat Gland Diseases; Skin Diseases, Bacterial; Hidradenitis; Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Tibulizumab Dose A (Experimental): Subcutaneous injection
  Interventions: Biological: Tibulizumab Dose A
- Tibulizumab Dose B (Experimental): Subcutaneous injection
  Interventions: Biological: Tibulizumab Dose B
- Placebo (Placebo Comparator): Subcutaneous injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Tibulizumab Dose A — Anti BAFF/IL-17 antibody. ZB-106
  Arms: Tibulizumab Dose A
Biological: Tibulizumab Dose B — Anti BAFF/IL-17 antibody. ZB-106
  Arms: Tibulizumab Dose B
Other: Placebo — ZB-106 Placebo
  Arms: Placebo

SUMMARY:
The study is a Phase 2, multi-center, randomized, double-blind, placebo-controlled study to evaluate the effects of tibulizumab over 16 weeks (Period 1) in adults with hidradenitis suppurativa, followed by a 16-week open-label extension period in which all participants will receive tibulizumab (Period 2)

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 70 years of age
* ≥6-month history of Hidradenitis suppurativa (HS)
* Total AN (abscess and inflammatory nodule) count ≥5
* HS lesions in ≥2 distinct anatomical areas, at least one of which is Hurley Stage II or III

Exclusion Criteria:

* Draining tunnel count >20
* Presence of another inflammatory condition or a skin condition that may interfere with study assessments
* Known to have immune deficiency or is immunocompromised
* Evidence or suspicion of active or latent tuberculosis
* History of opportunistic, chronic, or recurrent infection requiring chronic antibiotic use, serious or life-threatening infection within 2 months, or had an infection requiring systemic antibiotics within 2 weeks
* Has active systemic candidiasis
* Unable to tolerate subcutaneous drug administration

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
[Period 1] Percent change from baseline in abscess and inflammatory nodule (AN) count at 16 weeks | Week 16
  AN count is calculated based on the sum of the abscesses and inflammatory nodules across different anatomical areas

SECONDARY OUTCOMES:
[Period 1] Achieving HiSCR50 at Week 16 | Week 16
  HiSCRO50 is defined as at least a 50% decrease in total abscess and inflammatory nodule (AN) count with no increase from baseline in abscess and/or draining fistula count
[Period 1] Achieving HiSCR75 at Week 16 | Week 16
  HiSCR75 is defined as at least a 75% decreased in total abscess and inflammatory nodule (AN) count with no increase from baseline in abscess and/or draining fistula count
[Period 1] Absolute change from baseline in Dermatology Life Quality Index (DLQI) score at Week 16 | Week 16
  The DLQI is a validated general dermatology questionnaire that consists of 10 items that assess subject health-related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). Each item uses a scale from 0 (not at all) to 3 (very much), with a total score being the sum of each question. The higher the total score the more a patient's life is affected by their skin condition.
[Period 1] Absolute change from baseline in Patient's Global Assessment of Hidradenitis Suppurativa (HS-PtGA) score at Week 16 | Week 16
  The HS-PtGA is a single item measure that asks the individual to rate the overall impact of HS on their quality of life, capturing their comprehensive perception of disease severity and treatment response.
[Period 1] Absolute change from baseline in Skin Pain Numeric Rating Scale (NRS) at Week 16 | Week 16
  The Skin Pain NRS is a single-item measure in which the participant rates the worst level of skin pain in the previous 24 hours on a scale from 0 (no pain) to 10 (worst pain imaginable).
[Period 1] Safety and tolerability of tibulizumab | Week 16
  Assessed by the incidence of all treatment-emergent adverse events (TEAEs), as well as changes from baseline in vital signs, electrocardiogram (ECG) parameters, and laboratory results.

CONTACTS AND LOCATIONS:
Locations (56):
- United States (31):
  - Medical Dermatology Specialists (Phoenix), Phoenix, Arizona
  - First OC Dermatology Research, Inc., Irvine, California
  - Wallace Medical Group, Inc., Los Angeles, California
  - Northridge Clinical Trials, Northridge, California
  - NorCal Clinical Research, Rocklin, California
  - Florida Academic Dermatology Center, Coral Gables, Florida
  - Georgia Skin & Cancer Clinic, Savannah, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Equity Medical LLC (Kentucky), Bowling Green, Kentucky
  - DS Research of Kentucky, LLC, Louisville, Kentucky
  - DelRicht LLC, Baton Rouge, Louisiana
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Skin Cancer and Dermatology Institute, Reno, Nevada
  - Equity Medical, New York, New York
  - OptiSkin Medical, New York, New York
  - Optima Research, Boardman, Ohio
  - ClinOhio Research Services, Columbus, Ohio
  - Apex Clinical Research Center, Mayfield Heights, Ohio
  - Best Skin Research LLC, Camp Hill, Pennsylvania
  - Palmetto Clinical Trial Services, Anderson, South Carolina
  - DelRicht Research, Mt. Pleasant, South Carolina
  - International Clinical Research - Tennessee LLC, Murfreesboro, Tennessee
  - BRCR Global Texas, Katy, Texas
  - DelRicht Research, Prosper, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Frontier Dermatology, Mill Creek, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Dermatology Specialists of Spokane, Spokane, Washington
- Canada (5):
  - Ryan Clinical Research Inc., Newmarket, Ontario
  - North York Research Inc, North York, Ontario
  - York Dermatology Clinic & Research Centre, Richmond Hill, Ontario
  - Centre de recherche Saint-Louis, Québec, Quebec
  - Saskatoon Dermatology Centre, Saskatoon, Saskatchewan
- Germany (7):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Klinikum Darmstadt, Darmstadt
  - University Hospital Dresden, Dresden
  - Versorgungsforschung in der Dermatologie und bei Pflegeberufen (IVDP), Hamburg
  - University Clinic Dermatology Heidelberg, Heidelberg
  - Klinik und Poliklinik für Dermatologie und Allergologie, München
  - University Hospital Muenster - Münster, Münster
- Hungary (2):
  - Semmelweis University, Budapest
  - University of Debrecen, Debrecen
- Poland (7):
  - RENEW Clinic, Bialystok
  - Provita Centrum Medyczne Sp. z o.o. Katowice, Katowice
  - Provita Sp. z o. o., Katowice
  - Centrum Badawcze Panaceum Agnieszka Brzezicka, Magdalena Lenkiewicz Sp z .o.o, Malbork
  - SOLUMED, Poznan
  - Laser Clinic S.C., Szczecin
  - Manufaktura Zdrowia i Urody, Warsaw
- Spain (4):
  - Edificio IMIBIC, Reina Sofia University Hospital, Córdoba
  - Gregorio Marañón General University Hospital, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No